CLINICAL TRIAL: NCT05485987
Title: An Open-Label Study to Evaluate Pharmacokinetics, Safety, and Efficacy of Vatiquinone in Children With Friedreich Ataxia Younger Than 7 Years of Age
Brief Title: A Study of Vatiquinone for the Treatment of Participants With Friedreich Ataxia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC743-NEU-005-FA
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia | interventions — alpha-tocotrienol quinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vatiquinone (Experimental): Participants will receive an oral solution (100 milligrams [mg]/milliliter [mL]) of vatiquinone (15 mg/kilogram [kg] if body weight <13 kg and 200 mg if body weight ≥13 kg) 3 times a day (TID) for 72 weeks.
  Interventions: Drug: Vatiquinone

INTERVENTIONS:
Drug: Vatiquinone — Vatiquinone will be administered per dose and schedule specified in the arm.
  Other Names: PTC743; EPI-743

SUMMARY:
The primary objective of the study is to assess the pharmacokinetics (PK) and safety of vatiquinone administered in participants with Friedreich ataxia (FA) younger than 7 years.

ELIGIBILITY:
Inclusion Criteria:

* Friedreich ataxia diagnosis (homozygous for GAA repeat expansion in intron-1 of FXN gene), confirmed by clinical genetic testing.
* Must be able to abstain from anticoagulants and any aspirin (including 81 mg) for 30 days before the Baseline Visit and for the duration of the study; any possible discontinuation of anticoagulants should be monitored and indicated by a specialist (for example, cardiologist, neurologist, or hematologist), and discontinuation will be noted by the prescribing physician.
* Must be able to abstain from strong cytochrome P450 (CYP) 3A4 inducers/inhibitors (for example, ketoconazole, rifampin, St. John's wort, grapefruit juice, or any grapefruit product) for at least 30 days prior to enrollment and for the duration of the study.
* Must be able to take vatiquinone oral solution with food.

Exclusion Criteria:

* Previous treatment with vatiquinone.
* Allergy to vatiquinone or sesame oil.
* Ejection fraction <50%.
* Participation in any other interventional clinical trial or receipt of any study drug in any other clinical trial within 60 days prior to the Baseline Visit. Participants may be rescreened after the exclusionary period of 60 days has passed.
* Concomitant use of interventional CoQ10, vitamin E, or any approved or non-approved medication for FA within 30 days prior to the Baseline Visit. These prohibited medications can be discontinued at the Screening Visit.

Note: Other inclusion and exclusion criteria may apply.

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
Plasma Concentration of Vatiquinone | Pre-morning dose (0 hour) at Week 4; 1 to 3 hours and 3 to 6 hours post-morning dose at Weeks 4, 12, and 24
Area Under the Curve (AUC) of Vatiquinone | Pre-morning dose (0 hour) at Week 4; 1 to 3 hours and 3 to 6 hours post-morning dose at Weeks 4, 12, and 24
Number of Participants With Adverse Events | Baseline up to Week 76

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States